CLINICAL TRIAL: NCT06785454
Title: A Phase 2, Multicenter, Randomized, Double Blind, Placebo Controlled, Crossover Study to Evaluate the Efficacy and Safety of Lorundrostat in Participants With Moderate to Severe Obstructive Sleep Apnea and Hypertension
Brief Title: A Study to Assess the Efficacy and Safety of Lorundrostat in Participants With Obstructive Sleep Apnea and Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mineralys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MLS-101-207
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: Blood Pressure; Hypertension; Hypertensive; Sleep Apnea; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Lorundrostat then Placebo (Experimental)
  Interventions: Drug: Lorundrostat; Drug: Placebo
- Sequence 2: Placebo then Lorundrostat (Experimental)
  Interventions: Drug: Lorundrostat; Drug: Placebo

INTERVENTIONS:
Drug: Lorundrostat — Lorundrostat tablet.
Drug: Placebo — Lorundrostat matching placebo tablet.

SUMMARY:
The primary purpose of the study is to assess the effect of lorundrostat taken orally (po) once a day on the Apnea-Hypopnea Index (AHI) in participants with moderate to severe obstructive sleep apnea (OSA) and hypertension.

DETAILED DESCRIPTION:
The study is a randomized, double-blind (DB), placebo controlled, crossover study. A 4-week screening period is followed by two DB 4-week treatment periods separated by a 2-week washout period. Participants must be 18 to 75 years old with moderate to severe OSA, hypertension and meet all applicable eligibility criteria. Participants who are medically prescribed and deemed compliant with positive airway pressure (PAP) therapy for greater than or equal to (>=) 4 hours per night (Continuous PAP [CPAP], or automatic PAP [autoPAP]) and for at least 3 months prior to the study enrollment are eligible for the study. Participants on PAP therapy should comply with PAP therapy for the duration of the study. Participants who are not currently on PAP therapy and not anticipated to start PAP for the duration of the study, are also eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 27 kilograms per meter square (kg/m^2)
2. Previously diagnosed with moderate-to-severe OSA
3. AHI ≥15 events per hour (/hr) prior to Randomization
4. AOBP SBP of ≥130 and less than or equal to (≤) 180 millimeter of mercury (mmHg) and AOBP diastolic blood pressure (DBP) ≥60 and ≤110 mmHg
5. Participants on CPAP or PAP therapy are eligible provided they are on PAP for ≥4 hours per night (documented) and for at least 3 months prior to the study enrollment (documented)
6. Participants not currently on PAP therapy, and not anticipated to start PAP for the duration of the study
7. Fertile male and female participants of childbearing potential, and their partners, must agree to use protocol-defined methods of highly effective contraception from the Screening Visit until 28 days after the last dose of study drug

Exclusion Criteria:

1. Type 2 diabetes mellitus (T2DM) with a glycosylated hemoglobin (HbA1c) greater than (>) 9 percent (%) (>74.9 millimoles per mol [mmol/mol]) at the Screening Visit or history of diabetic ketoacidosis in the 6 months prior to the Screening Visit
2. Participants on a glucagon-like peptide-1 (GLP-1) agonist.
3. Any surgery for sleep apnea or major ear, nose or throat surgery, including tonsillectomy and adenoidectomy within 3 months prior to Screening, or planned during participation in the study or within 1 month of the last study visit.
4. Have diagnosis of central or mixed sleep apnea with % of mixed or central apneas/hypopneas ≥50%, or diagnosis of Cheyne Stokes Respiration
5. Diagnosis of Obesity Hypoventilation Syndrome or daytime hypercapnia
6. Use of bilevel positive airway pressure (BiPAP) therapy.
7. eGFR less than (<) 45 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) at Screening using serum creatinine or cystatin-C
8. History of clinically relevant medical, behavioral, or psychiatric disorder, other than OSA, that is associated with insomnia or excessive sleepiness
9. Diagnosed with Child-Pugh Class C
10. Participants who regularly use caffeine stimulants or participants who are unwilling to reduce intake to 300 mg per day (approximately 3 cups of coffee), for a period of at least 3 days prior to the Screening visit or a sleep study
11. Treatment with MRAs and/or epithelial sodium channel (ENaC) inhibitors within 1 month of the Screening Visit
12. Requirement for nocturnal use of supplemental oxygen
13. Women who are pregnant, plan to become pregnant, or are breastfeeding
14. Unstable or currently symptomatic cardiovascular disease or hospitalization in the 6 months prior to Screening
15. Previously diagnosed, recurrent orthostatic hypotension
16. Current night-shift worker or anticipated to become a night-shift worker for 3 days continuously during the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Placebo-adjusted Change From Baseline in AHI at Week 4 | Baseline, Week 4

SECONDARY OUTCOMES:
Placebo-adjusted Change From Baseline in Nighttime Average Systolic Blood Pressure (SBP) at Week 4 | Baseline, Week 4
Placebo-adjusted Change From Baseline in Automated Office Blood Pressure (AOBP) SBP at Week 4 | Baseline, Week 4
Placebo-adjusted Change From Baseline in Functional Outcomes of Sleep Questionnaire-10 (FOSQ-10) at Week 4 | Baseline, Week 4
Placebo-adjusted Change From Baseline in Epworth Sleepiness Scale (ESS) at Week 4 | Baseline, Week 4
Placebo-adjusted Change From Baseline in Patient-Reported Outcomes Measurement Information System - Sleep Disturbance (PROMIS-SD) at Week 4 | Baseline, Week 4
Placebo-adjusted Change From Baseline in PROMIS Sleep-Related Impairment (SRI) at Week 4 | Baseline, Week 4

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - The University of Alabama, Tuscaloosa, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Preferred Research Partners Inc., Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - The Neurology Center of Southern California - Profound Research, LLC, Carlsbad, California
  - Probe Clinical Research Corporation, Riverside, California
  - Research Carolina Elite, Denver, Colorado
  - Nouvelle Clinical Research, Cutler Bay, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - CNS Healthcare - Orlando (Clinical Neuroscience Solutions), Orlando, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Centricity Research Rincon Pulmonology, Rincon, Georgia
  - Chicago Research Center Inc, Chicago, Illinois
  - Centennial Medical Group, Columbia, Maryland
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Henry Ford Health System/Henry Ford Medical Center - Columbus, Novi, Michigan
  - Revive Research Institute, Inc, Southfield, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Patient First MD, Middletown, New Jersey
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Northwest Research Center, Portland, Oregon
  - CNS Healthcare - Memphis (Clinical Neuroscience Solutions - Memphis), Memphis, Tennessee
  - Huntsville Research Institute LLC, Huntsville, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No